CLINICAL TRIAL: NCT03412695
Title: Development of a Decision Support System to Prevent and Treat Disease-related Malnutrition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: University of Oslo (Other)
Responsible Party: Principal Investigator, Mari Mohn Paulsen, Project coordinator, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2016/1464
Record Dates: First submitted 2018-01-10; First posted 2018-01-26 (Actual); Last update posted 2019-07-31 (Actual); Status verified 2019-07

CONDITIONS: Malnutrition
Keywords: Disease-related malnutrition; eHealth; Decision support system; Clinical nutrition
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): Use of the MyFood tool among patients and nurses (intervention group)
  Interventions: Device: MyFood
- Arm B (No Intervention): No intervention. Regular hospital routines

INTERVENTIONS:
Device: MyFood — Patients included in the intervention group will use the MyFood app to record their dietary intake. Nurses will use the report and recommendations in the MyFood tool to follow up the nutritional treatment of the patients.
  Arms: Arm A

SUMMARY:
The prevalence of disease-related malnutrition among hospitalized patients is 30-50%. There is a lack of tools to follow up the nutritional treatment of these patients. The investigators develop the decision support system "MyFood" which can be used to assess patients' dietary intake, evaluate intake against individual needs, and propose nutrition related measures and an individual nutrition plan for each patient. The investigators will study the clinical effects of using MyFood among hospitalized patients. In addition the implementation of the tool among healthcare workers will be studied.

DETAILED DESCRIPTION:
The prevalence of disease-related malnutrition among hospitalized patients is 30-50%. Disease-related malnutrition increase the morbidity and mortality among patients and leads to longer length of stay. There is a lack of tools to follow up the nutritional treatment of patients at nutritional risk. The decision support system "MyFood" is developed in the project with the purpose to prevent and treat disease-related malnutrition. MyFood includes 4 modules: 1) A function to register patient needs and symptoms, 2) Dietary assessment function, 3) Automatic evaluation of dietary intake compared to individual needs, 4) Feedback, including a report on intake of energy, protein, and liquids compared to individual needs, and recommendations for nutritional measures and an individual nutrition plan.

Clinical effects of using MyFood among hospitalized patients will be studied in a randomized controlled trial. In addition, the implementation of the tool among nurses and other healthcare workers will be explored.

ELIGIBILITY:
Exclusion Criteria:

* <72 hours expected hospital stay
* Terminal patients
* Pregnant
* Psychiatric patients
* Patients who cannot read the Norwegian Language
* Patients diagnosed with: sickle cell anemia, haemophilia, or deep vein thrombosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-08-22 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
Change in body weight (kg) during hospital stay | 2 times each week, from patient admission (day 1) to hospital discharge (on average day 11)
  Measured standing on an electronic scale

SECONDARY OUTCOMES:
Patient length of hospital stay | At the day of patient discharge (on day 11)
  Length of hospital stay (LOS) will be measured for all participating patients. Average LOS in the intervention group will be compared with the average LOS in the control group
Change in body Composition | 2 times each week, from patient admission (day 1) to hospital discharge (on average day 11)
  Fat free mass, muscle mass, fat mass, and phase angle. Measured by bioelectrical impedance analysis.
Proportion of patients who receives a nutrition diagnose | Assessed from medical journals every second day during each patient's hospital stay (11 days on average)
  Number of patients who receives a nutrition diagnose (E46.00) will be measured among patients participating in the study. Proportion of patients who receives a nutrition diagnose in the intervention group will be compared with the proportion of patients who receives a nutrition diagnose in the control group.
Proportion of patients who get implemented nutrition-related measures | Assessed from medical journals every second day during each patient's hospital stay (11 days on average)
  The decision support system gives recommendations for nutritional-related measures, based on individual symptoms and dietary intake compared to needs.
Proportion of patients who receive a nutrition plan | Assessed from the participating patients' medical journals on day 2 and every second day during hospital stay (11 days on average)
  According to the national guidelines all patients at nutritional risk should have an individual nutrition plan. The decision support system will generate a suggested nutrition plan, based on information recorded in the system. Proportion of patients in the intervention group who receives a nutrition plan, compared to proportion in the control group will be measured
Re-admissions | 30 days after discharge
  Unplanned re-admissions
Patient generated subjective global assessment (PG-SGA) score | Measured on day 1 and at admission (day 11 on average)
  The patient generated subjective global assessment (PG-SGA) is a form including questions on weight development, food intake, symptoms, and activity level and function

CONTACTS AND LOCATIONS:
Locations (1):
- Oslo university hospital, Rikshospitalet, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Paulsen MM, Varsi C, Andersen LF. Process evaluation of the implementation of a decision support system to prevent and treat disease-related malnutrition in a hospital setting. BMC Health Serv Res. 2021 Mar 25;21(1):281. doi: 10.1186/s12913-021-06236-3. PMID 33766017
- [Derived] Paulsen MM, Paur I, Gjestland J, Henriksen C, Varsi C, Tangvik RJ, Andersen LF. Effects of using the MyFood decision support system on hospitalized patients' nutritional status and treatment: A randomized controlled trial. Clin Nutr. 2020 Dec;39(12):3607-3617. doi: 10.1016/j.clnu.2020.03.012. Epub 2020 Mar 19. PMID 32241711